CLINICAL TRIAL: NCT06670781
Title: Standardized Goal-Directed vs. Self-Directed Valsalva Maneuver for the Assessment of Patent Foramen Ovale
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: OHSN CRRF ID - 6016
Record Dates: First submitted 2024-10-24; First posted 2024-11-01 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-09

CONDITIONS: Stroke
Keywords: Bubble study; Stroke; Echocardiography; patent foramen ovale
MeSH Terms: conditions — Stroke; Foramen Ovale, Patent

STUDY DESIGN:
Intervention Model Description: A blinded comparative crossover diagnostic accuracy study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control - standard of care: Self-Directed Valsalva maneuver (Sham Comparator): The Valsalva maneuver is performed by the patient taking a normal (or deep) inspiration, followed by forceful expiration against a closed airway for up to 15 to 20 sec and then release of the expiratory effort on entry of saline into the right atrium.
  Interventions: Device: Experimental: Intervention arm: Goal-Directed Valsalva maneuver; Device: Control - standard of care: Self-Directed Valsalva maneuver
- Intervention arm: Goal-Directed Valsalva maneuver (Active Comparator): For the Goal directed Valsalva maneuver, the same method patients are instructed to blow into a plastic pipe connected to the manometer device, in order to reach a pressure of 40 mmHg for at least 5 seconds. Then patients are instructed to exhale quickly.
  Interventions: Device: Experimental: Intervention arm: Goal-Directed Valsalva maneuver; Device: Control - standard of care: Self-Directed Valsalva maneuver

INTERVENTIONS:
Device: Experimental: Intervention arm: Goal-Directed Valsalva maneuver — For the Goal directed Valsalva maneuver, the same method patients are instructed to blow into a plastic pipe connected to the manometer device, in order to reach a pressure of 40 mmHg for at least 5 seconds. Then patients are instructed to exhale quickly.
Device: Control - standard of care: Self-Directed Valsalva maneuver — The Valsalva maneuver is performed by the patient taking a normal (or deep) inspiration, followed by forceful expiration against a closed airway for up to 15 to 20 sec and then release of the expiratory effort on entry of saline into the right atrium.

SUMMARY:
Ischemic stroke represents a major public health issue, leading to significant disabilities and deaths worldwide. When no clear cause for stroke is found following a comprehensive cardiovascular evaluation (no atrial fibrillation, cardiac masses, or atherosclerosis) i.e. cryptogenic stroke, it is recommended to search for a patent foramen ovale (PFO), especially in young patients. It is estimated that cryptogenic stroke accounts for 30% to 40% of ischemic strokes. Transthoracic echocardiography (TTE) with bubble study at rest and during Valsalva maneuver is the reference method for the diagnosis of PFO. The treatment of PFO using a closure device has demonstrated a significant reduction in recurrent stroke events in patients with PFO and cryptogenic stroke. The Valsalva maneuver is currently achieved using self-directed maneuver i.e. patients are instructed to ''bear down'' or ''strain as if attempting to move your bowels.'' These instructions are subjective and depend largely on individuals understanding and effort. A Goal-Directed Valsalva Maneuver using a manometer has been shown to be a more reproducible way to perform the Valsalva achieving more sensitivity in different settings such as hypertrophic cardiomyopathy but its incremental diagnostic value for the detection of PFO has not been yet evaluated.

The aim of the present study is to compare the sensibility and specificity of two methods of Valsalva maneuver for the detection of PFO. We hypothesize that Goal-Directed Valsalva Maneuver will significantly increase the detection rate of PFO compared to Self-Directed Valsalva Maneuver.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for a clinically indicated TTE and bubble study

Exclusion Criteria:

* Inability to provide informed consent
* Inability to insert an IV line
* Inability to perform a Self-Directed Valsalva maneuver
* Patient wishing to keep his mask on

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Rate of detection of PFO by Self-Directed Valsalva Maneuver and Goal-Directed Valsalva Maneuver. | From enrollment to the end of echocardiogram (40 minutes from enrollment).

SECONDARY OUTCOMES:
Rate of large shunt positive bubble study. | From enrollment to the end of echocardiogram (40 minutes from enrollment).
Rate of detection of PFO by Self-Directed Valsalva Maneuver and Goal-Directed Valsalva Maneuver in women and in men. | From enrollment to the end of echocardiogram (40 minutes from enrollment).

CONTACTS AND LOCATIONS:
Overall Officials: Dr. David Messika-Zeitoun, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bernard S, Churchill TW, Namasivayam M, Bertrand PB. Agitated Saline Contrast Echocardiography in the Identification of Intra- and Extracardiac Shunts: Connecting the Dots. J Am Soc Echocardiogr. 2020 Oct 23:S0894-7317(20)30615-5. doi: 10.1016/j.echo.2020.09.013. Online ahead of print. PMID 34756394
- [Background] Zhao E, Du Y, Xie H, Zhang Y. Modified Method of Contrast Transthoracic Echocardiography for the Diagnosis of Patent Foramen Ovale. Biomed Res Int. 2019 May 9;2019:9828539. doi: 10.1155/2019/9828539. eCollection 2019. PMID 31211145
- [Background] Mas JL, Derumeaux G, Guillon B, Massardier E, Hosseini H, Mechtouff L, Arquizan C, Bejot Y, Vuillier F, Detante O, Guidoux C, Canaple S, Vaduva C, Dequatre-Ponchelle N, Sibon I, Garnier P, Ferrier A, Timsit S, Robinet-Borgomano E, Sablot D, Lacour JC, Zuber M, Favrole P, Pinel JF, Apoil M, Reiner P, Lefebvre C, Guerin P, Piot C, Rossi R, Dubois-Rande JL, Eicher JC, Meneveau N, Lusson JR, Bertrand B, Schleich JM, Godart F, Thambo JB, Leborgne L, Michel P, Pierard L, Turc G, Barthelet M, Charles-Nelson A, Weimar C, Moulin T, Juliard JM, Chatellier G; CLOSE Investigators. Patent Foramen Ovale Closure or Anticoagulation vs. Antiplatelets after Stroke. N Engl J Med. 2017 Sep 14;377(11):1011-1021. doi: 10.1056/NEJMoa1705915. PMID 28902593
- [Background] Mojadidi MK, Winoker JS, Roberts SC, Msaouel P, Zaman MO, Gevorgyan R, Tobis JM. Accuracy of conventional transthoracic echocardiography for the diagnosis of intracardiac right-to-left shunt: a meta-analysis of prospective studies. Echocardiography. 2014 Oct;31(9):1036-48. doi: 10.1111/echo.12583. Epub 2014 Apr 2. PMID 24689727
- [Background] Saric M, Armour AC, Arnaout MS, Chaudhry FA, Grimm RA, Kronzon I, Landeck BF, Maganti K, Michelena HI, Tolstrup K. Guidelines for the Use of Echocardiography in the Evaluation of a Cardiac Source of Embolism. J Am Soc Echocardiogr. 2016 Jan;29(1):1-42. doi: 10.1016/j.echo.2015.09.011. PMID 26765302
- [Background] Cohen A, Donal E, Delgado V, Pepi M, Tsang T, Gerber B, Soulat-Dufour L, Habib G, Lancellotti P, Evangelista A, Cujec B, Fine N, Andrade MJ, Sprynger M, Dweck M, Edvardsen T, Popescu BA; Reviewers: This document was reviewed by members of the 2018-2020 EACVI Scientific Documents Committee; chair of the 2018-2020 EACVI Scientific Documents Committee. EACVI recommendations on cardiovascular imaging for the detection of embolic sources: endorsed by the Canadian Society of Echocardiography. Eur Heart J Cardiovasc Imaging. 2021 May 10;22(6):e24-e57. doi: 10.1093/ehjci/jeab008. PMID 33709114
- [Background] Yaghi S, Bernstein RA, Passman R, Okin PM, Furie KL. Cryptogenic Stroke: Research and Practice. Circ Res. 2017 Feb 3;120(3):527-540. doi: 10.1161/CIRCRESAHA.116.308447. PMID 28154102
- [Background] Mojadidi MK, Mahmoud AN, Patel NK, Elgendy IY, Meier B. Cryptogenic Stroke and Patent Foramen Ovale: Ready for Prime Time? J Am Coll Cardiol. 2018 Sep 4;72(10):1183-1185. doi: 10.1016/j.jacc.2018.03.549. No abstract available. PMID 30165998